CLINICAL TRIAL: NCT00437827
Title: A Multicenter, Randomized, Blinded, Controlled, Parallel Group Trial to Demonstrate the Efficacy of rEEG Guided Pharmacotherapy of Subjects With Depression Treatment Failure
Brief Title: rEEG Guided Pharmacotherapy of Subjects With Depression Treatment Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MYnd Analytics (Industry)
Responsible Party: Daniel Hoffman, MD, Chief Medical Officer, CNS Response, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rEEGTRD010; CNSR #010
Record Dates: First submitted 2007-01-17; First posted 2007-02-21 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Each subject in this arm will receive depression therapy similar to that used by the Star*D study - a major depression study conducted in the United States (Sequenced Treatment Alternatives to Relieve Depression (STAR*D) trial. Am J Psychiatry 2006; 163:1905-1917)
  Interventions: Other: Star*D algorithm
- 2 (Experimental): Each subject in this arm will receive therapy based upon an individualized rEEG report which provides one or more treatment options with the highest probability of success.
  Interventions: Other: rEEG-guided therapy

INTERVENTIONS:
Other: Star*D algorithm — Standard of care based upon the therapies selected in the Star*D study.
  Other Names: Standard of Care
  Arms: 1
Other: rEEG-guided therapy — An rEEG report is based upon a process that utilizes a patient's drug-free QEEG to predict successful treatment strategies.
  Other Names: EEG-based technology
  Arms: 2

SUMMARY:
This study is testing a process (rEEG)for selecting the most appropriate medication(s) to treat a patient's depression versus a control group being treated according to a standardized method, the modified Star*D Algorithm. Qualified subjects will be randomized to the experimental (rEEG guided) group, or the control group and treated for 12 weeks. Medications utilized in this study are currently marketed. All visits, physical exam, rEEG, labs, rating scales and medications are provided at no cost to the patient.

DETAILED DESCRIPTION:
This study is testing a process (rEEG)for selecting the most appropriate medication(s) to treat a patient's depression versus a control group being treated according to a standardized method, the modified Star*D Algorithm. Qualified subjects will be randomized to the experimental (rEEG guided) group, or the control group and treated for 10 weeks. Medications utilized in this study are currently marketed. All visits, physical exam, rEEG, labs, rating scales and medications are provided at no cost to the patient.

To qualify for entry into the study, patients must be:

1. 18 years of age or older.
2. Diagnosis of Major Depressive Disorder. Subjects may meet criteria for both melancholic and atypical depression.
3. Have failed 1 or more SSRIs, or have failed 2 or more antidepressants in at least 2 drug classes.

And patients must not have:

1. History of: closed head injury with unconsciousness, craniotomy, cerebral metastases, cerebrovascular accident; no current diagnosis of seizure disorder, bipolar disorder, schizophrenia, dementia, mental retardation, substance abuse, or major depression with psychotic features; or use of depot neuroleptics in last 12 months.
2. Known pregnancy and/or lactation, or intent to become pregnant during this study.

Medications that can be used in this study are:

Anti-depressants: fluoxetine, sertraline, paroxetine, desipramine, imipramine, nortriptyline,amitriptyline, clomipramine, bupropion, venlafaxine

Stimulants & MAO Inhibitors: moclobemide, tranylcypromine, selegiline, methylphenidate, dextroamphetamine, dexlevoamphetamine, pemoline, lamotrigine, topiramate

Benzodiazepines: lorazepam, clonazepam, alprazolam

Anti-convulsants: carbamazepine, lithium, divalproex, gabapentin

Beta Blockers: metoprolol, propranolol, atenolol

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Diagnosis of Major Depressive Disorder validated by SCID. Subjects may meet criteria for both melancholic and atypical depression per this protocol.
3. Have failed three or more antidepressant regimens during the current depressive episode with minimum daily dose(s) as defined in the Medication History for Depression Case Report Form and for a minimum duration of treatment of at least 4 weeks. For purposes of the Study, augmentation will be considered a separate regimen.
4. Able to stop all medications for 5 half-lives of the medication(s), with the exception of hormones, thyroid, hydrochlorthiazide and Ambien. See Appendix II for a list of the half-lives of medications.

Exclusion Criteria:

1. History of: closed head injury with unconsciousness, craniotomy, cerebral metastases, cerebrovascular accident; no current diagnosis of seizure disorder, bipolar disorder, schizophrenia, dementia, mental retardation, substance abuse, or major depression with psychotic features; or use of depot neuroleptics in last 12 months.
2. Participation in any other therapeutic drug study evaluating a treatment for depression within 60 days preceding inclusion, unless drug(s) half-life is known.
3. Known pregnancy and/or lactation, or intent to become pregnant during this study.
4. Doesn't qualify via rEEG analysis due to:

   * Potential physiologic abnormality
   * Low abnormality in comparison to current rEEG database
   * No strong prediction by rEEG analysis for any particular medication class

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Two group comparison of QIDS-SR16 and Q-LES-Q-SF | after 12 weeks of treatment

SECONDARY OUTCOMES:
Two group comparison of MADRS, Clinical Global Improvement and Severity. | after 12 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Charles DeBattista, MD, Principal Investigator — Stanford University; Gustavo Kinrys, M.D., Principal Investigator — Cambridge Hospital; Steven G Potkin, MD, Principal Investigator — University of California, Irvine; Daniel Hoffman, MD, Study Chair — MYnd Analytics
Locations (13):
- United States (13):
  - Behavioral Research Specialists, Glendale, California
  - University of California - Irvine, Irvine, California
  - Shanti Research and Clinical Trials, San Bernardino, California
  - Stanford University, Stanford, California
  - Elite Clinical Trials, Wildomar, California
  - Radiant Research, Denver, Colorado
  - Hawaii Clinical Research Center, Honolulu, Hawaii
  - Rush University, Chicago, Illinois
  - McClean Hospital/Harvard, Belmont, Massachusetts
  - Harvard Medical School - Cambridge Hospital, Cambridge, Massachusetts
  - Alpha Behavioral Care, P.A., Summit, New Jersey
  - Cornell University, New York, New York
  - Univ of TX Health Science Center, San Antonio, Texas